CLINICAL TRIAL: NCT05350930
Title: Multidisciplinary Care Program to Secure MEdication Therapy for HematoLOgy Patients Receiving Injectable Anticancer Drugs
Acronym: Melodia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0292
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chemotherapy Effect; G-CHOP Chemotherapy; R-CHOP Chemotherapy
Keywords: Haematology; Pharmaceutical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- R-CHOP or G-CHOP chemotherapy: Patients with hematological malignancies receiving R-CHOP or G-CHOP chemotherapy
  Interventions: Other: Assessment of patient satisfaction regarding tele-consultation; Other: Literacy questionnaire; Other: Collection of socio-demographic characteristics; Other: Assessment of patient knowledge on chemotherapy side effects and support medications; Other: Assessment of patient satisfaction on pharmaceutical follow-up

INTERVENTIONS:
Other: Assessment of patient satisfaction regarding tele-consultation — Questionnaire completed following the teleconsultation, if applicable.
Other: Literacy questionnaire — Questionnaire completed during hospitalization for the first chemotherapy cycle
Other: Collection of socio-demographic characteristics — Questionnaire completed during patient hospitalization for the first chemotherapy cycle
Other: Assessment of patient knowledge on chemotherapy side effects and support medications — Questionnaire completed during patient hospitalization for the first, second and sixth cycle of chemotherapy
Other: Assessment of patient satisfaction on pharmaceutical follow-up — Questionnaire completed during patient hospitalization for the sixth chemotherapy cycle

SUMMARY:
Several experiences of multidisciplinary care pathways associating oncologists, pharmacists and nurses have been reported for cancer patients, with positive results on medication management safety, reduction of Drug-Related Problems (DRPs), and re-hospitalizations.

This study aims to evaluate the impact of a multidisciplinary city-hospital follow-up program on medication management safety in haematological oncology patients receiving intravenous chemotherapy in onco-haematology. Additional aspects will be evaluated, such as the impact of the follow-up on the city-hospital link, satisfaction of patients and professionals involved in the follow-up and the use of telecare

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18 years or older With hematological malignancy at any stage Initiating R-CHOP or G-CHOP chemotherapy Who do not object to participation in the study and use of collected data

Exclusion Criteria:

* Patients already enrolled in a clinical trial evaluating any drug product
* Patients living in an institution
* Patients protected by law

  * Adults subject to a legal protection measure (curatorship, guardianship) (article L1121-8 of the CSP)
  * Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care and persons admitted to a health or social establishment (article L1121-6 of the CSP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients treated in the hematology department of a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical impact of pharmacist interventions at first cycle of chemotherapy, according to the CLEO© scale. | 6 months after inclusion
  Each pharmacist intervention performed during patient follow-up will be rated according to its expected level of clinic impact (major, moderate, minor, null)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud - Hospices Civils de lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: Undecided